CLINICAL TRIAL: NCT01651871
Title: A Phase 2, Multicenter, Parallel-Group, Randomized, Double-Blind, Placebo- And Active Comparator-Controlled, Combination Study Of S-555739 And Cetirizine HCl In Adult Patients With Seasonal Allergic Rhinitis
Brief Title: Combination Study Of S-555739/Cetirizine HCl In Adult Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1210D1526
Record Dates: First submitted 2012-07-17; First posted 2012-07-27 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Agents, anti allergic; Nasal congestion; Sneezing; Nasal discharge; D prostanoid (DP) receptor antagonist
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Nasal Obstruction; Sneezing; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Treatment Group 1 (Experimental)
  Interventions: Drug: S-555739 Dose 1; Drug: Cetirizine HCl Dose 1
- Treatment Group 2 (Experimental)
  Interventions: Drug: S-555739 Dose 2; Drug: Cetirizine HCl Dose 1; Drug: S-555739 placebo
- Treatment Group 3 (Experimental)
  Interventions: Drug: S-555739 Dose 1; Drug: Cetirizine HCl placebo
- Treatment Group 4 (Active Comparator)
  Interventions: Drug: Cetirizine HCl Dose 1; Drug: S-555739 placebo
- Treatment Group 5 (Placebo Comparator)
  Interventions: Drug: S-555739 placebo; Drug: Cetirizine HCl placebo

INTERVENTIONS:
Drug: S-555739 Dose 1
  Arms: Treatment Group 1; Treatment Group 3
Drug: S-555739 Dose 2
  Arms: Treatment Group 2
Drug: Cetirizine HCl Dose 1
  Arms: Treatment Group 1; Treatment Group 2; Treatment Group 4
Drug: S-555739 placebo
  Arms: Treatment Group 2; Treatment Group 4; Treatment Group 5
Drug: Cetirizine HCl placebo
  Arms: Treatment Group 3; Treatment Group 5

SUMMARY:
The primary objective of the study was to examine the efficacy and safety of S-555739/cetirizine HCl compared with the individual components and placebo.

ELIGIBILITY:
Inclusion Criteria:

* History and diagnosis of seasonal allergic rhinitis by skin prick test
* Have nasal symptom scores as defined by the study protocol
* Able to comply with study procedures

Exclusion Criteria:

* Any nasal disease or abnormality, active respiratory tract infections within the past 2 weeks, or recent nasal surgery or sinus surgery at Screening
* Use of any prohibited concomitant drugs or therapies

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 779 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in average morning/evening (AM/PM) reflective Total Nasal Symptom Score (rTNSS) | Change from baseline through the 2-week treatment period (Day 2 through Day 15)
Incidence of adverse events (AEs) | From Screening period to Week 6 (Follow-up)

SECONDARY OUTCOMES:
Change in average AM/PM instantaneous Total Nasal Symptom Score (iTNSS) | Change from baseline through the 2-week treatment period (Day 2 through Day 15)
Change in average AM/PM Total Ocular Symptom Score | Change from baseline through the 2-week treatment period (Day 2 through Day 15)
Assessment of Quality of Life | Change from Week 3 to Week 5
Assessment of vital signs | At Week 1 (Screening), Week 2, Week 3, Week 4, and Week 5
Assessment of clinical laboratory parameters | At Week 1 (Screening), Week 4, Week 5, and Week 6 (Follow-up)
Assessment of electrocardiogram (ECG) findings | At Week 1 (Screening) and Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi